CLINICAL TRIAL: NCT03513835
Title: Diagnostic Screening Tests and Potential Biomarkers in Mitochondrial Myopathies
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, MD, PhD-student, Rigshospitalet, Denmark
Other Study IDs: H-17032512
Record Dates: First submitted 2018-01-15; First posted 2018-05-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Mitochondrial Myopathies; Healthy Controls
MeSH Terms: conditions — Mitochondrial Myopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mitochondrial myopathy
  Interventions: Diagnostic Test: Diagnostic screenings tests
- Healthy controls
  Interventions: Diagnostic Test: Diagnostic screenings tests

INTERVENTIONS:
Diagnostic Test: Diagnostic screenings tests — Handgrip test, 12-minute walk test and 6-minute walk test. Biomarkers: acyl-carnitine profile and GDF-15.

SUMMARY:
The purpose of this study is to develop simple diagnostic screeningtests and investigate potential biomarkers for identifying patients with abnormalities of mitochondrial function, which also can be used as outcome measures in future clinical trials. The study will investigate two submaximal tests: a submaximal handgrip test and a walking test. Furthermore investigators will investigate Acyl-carnitine profiles and GDF-15 levels in patients with mitochondrial myopathy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* verified mitochondrial myopathy
* or healthy control
* or disease control (another neuromuscular disease)

Exclusion Criteria:

* Patient has any prior or current medical conditions that, in the judgment of the Investigator, would prevent the patient from safely participating in and/or completing all study requirements.
* Patient has symptoms of mitochondrial myopathy due to known secondary mitochondrial dysfunction
* Patient does not have the cognitive capacity to understand/comprehend and complete all study assessments.
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Genetically verified primary Mitochondrial disorder with myopathy.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Serum lactate / pyruvate ratio | 1 hour
  Changes between: before, during and after submaximal exercise
Serum Acyl-carnitine levels | 1 hour
  Changes between: before and after exercise, fasted and fed.
Serum GDF-15 | 1 hour
  Changes between: before and after exercise, fasted and fed.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lokken N, Skriver SV, Khawajazada T, Storgaard JH, Vissing J. Plasma lactate responses during and after submaximal handgrip exercise are not diagnostically helpful in mitochondrial myopathy. Mitochondrion. 2021 Sep;60:21-26. doi: 10.1016/j.mito.2021.07.002. Epub 2021 Jul 15. PMID 34273558